CLINICAL TRIAL: NCT05065801
Title: Randomized Phase II Trial Evaluating the Efficacy of a Sequential Treatment Gemcitabine Plus Nab-paclitaxel (Gembrax) Followed by Folfirinox Versus Folfirinox Alone in Patients Treated in First Metastatic Line Pancreatic Cancer
Brief Title: Efficacy of Gembrax Followed by Folfirinox Versus Folfirinox Alone in First Metastatic Line Pancreatic Cancer Patients
Acronym: GABRINOX2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROICM 2021-02 GAB
Record Dates: First submitted 2021-09-20; First posted 2021-10-04 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: pancreatic; cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GEMBRAX/FOLFIRINOX Arm A (Experimental): One cycle:
  * D1, D8 and D15 GEMBRAX: Albumin bound paclitaxel 125mg / m² followed by Gemcitabine 1000mg / m² followed by 2 weeks of rest
  * D29 and D43 FOLFIRINOX: Oxaliplatin 85mg / m², Irinotecan 180mg / m², Folinic acid 400 mg / m², 5-fluorouracil 400mg / m² in bolus followed by continuous administration over 46h at 2400mg / m² followed by 2 weeks of rest.
  A maximum of 6 cycles (12 months) of chemotherapy will be administered to patients in arm A.
  Interventions: Combination Product: GEMBRAX/FOLFIRINOX Arm A
- FOLFIRINOX Arm B (Active Comparator): One cycle :
  D1, D15, D29 and D43 FOLFIRINOX: Oxaliplatin 85mg / m², Irinotecan 180mg / m², Folinic acid 400mg / m², 5-fluorouracil 400mg / m² as a bolus followed by continuous administration over 46h at 2.400mg / m² followed by 2 weeks of rest.
  A maximum of 3 cycles (6 months) of chemotherapy will be administered to patients in arm B.
  Interventions: Combination Product: FOLFIRINOX Arm B

INTERVENTIONS:
Combination Product: GEMBRAX/FOLFIRINOX Arm A — Patients in the experimental arm received sequential treatment: A maximum of 6 cycles (12 months) of chemotherapy; One cycle = 3 administrations of GEMBRAX followed by 2 administrations of FOLFIRINOX
  Arms: GEMBRAX/FOLFIRINOX Arm A
Combination Product: FOLFIRINOX Arm B — Patients in this arm received : A maximum of 3 cycles (6 months) of chemotherapy. One cycle = 4 administrations of FOLFIRINOX
  Arms: FOLFIRINOX Arm B

SUMMARY:
The aim of this study is to evaluate the efficacy of sequential treatment (Gabrinox) comprising Gembrax regimen (Gemcitabine -Abraxane) followed by the Folfirinox regimen (5FU, Oxaliplatin and Irinotecan) compared to folfirinox alone in patients treated in first metastatic line pancreatic cancer

DETAILED DESCRIPTION:
Pancreatic cancer is the third leading cause of cancer death in 2016, surpassing breast cancer. It is estimated that by 2030 pancreatic cancer will become the second leading cause of cancer death after lung cancer.

Its prognosis is very poor, with a 5-year overall survival rate (OS) at all stages of 5.5%.

In France, its incidence doubled in men and tripled in women between 1982 and 2012. The World Standardized Rate (MSR) for men and women respectively was 4.9% and 2% in 1980 and 10.2% and 6.9% in 2012. This means an annual rate of change of 2.3 for men to 3.9 for women.

Its diagnosis is often late, carried out in 50% of cases at stage 4, with limited treatment options, explaining its low survival rate at 5 years.

Until 2011, gemcitabine remained the only validated standard with a median survival of 6 months.

Many combinations with gemcitabine have been evaluated but have shown no significant survival advantage over Gemzar alone.

The most promising results reported to date remain the combination of oxaliplatin, irinotecan and 5 fluoro-uracil (FOLFIRINOX), which became the standard metastatic first-line treatment thanks to the results of the phase III study, ACCORD11, randomizing gemcitabine to FFX with for the first time, a significant gain in median survival, progression-free survival and response rate in favor of the experimental arm of 6.8 months vs. 11.1 months respectively ([HR 0.57, 95 % IC, 0.45-0.7 3];p<0.001), 3.3vs6.4 ([HR 0.47, 95 % IC, 0.37- 0.59];p<0.001) et de 9.4 % vs 31.6 % ; p>0.001.

In 2013, the combination gemcitabine nab-paclitaxel (GEMBRAX) showed, in a randomized phase III study, compared to gemcitabine, a significant gain in terms, median survival, survival without progression and response rate in favor of the experimental arm, respectively for gemcitabine vs GEMBRAX, 6.7 months vs 8.5 months ([HR 0.72, 95 % IC, 0.62-0.83];p<0.001) ; 3.7vs 5.5. ([HR 0.69, 95 % IC, 0.58- 0.82];p<0.001) et de 7 % vs 23% ; p>0.001.

FOLFIRINOX and GEMBRAX, two chemotherapy protocols which have shown their effectiveness in the 1st metastatic line with a gain in terms of response rate, progression-free survival and median survival but with increased grade 3/4 toxicities, compared to treatment with gemcitabine.

For FOLFIRINOX: a neutropenia rate of 45.7% vs 21% including 5.4% of febrile neutropenia vs 1.2, a rate of diarrhea of 12.7% vs 1.8% and peripheral neuropathies of 9% vs 0

For GEMBRAX neutropenia 38% VS 27% including 3% febrile neutropenia VS 1%, 6% diarrhea vs 1% and peripheral neuropathy 17% vs 1%:

Given the high toxicities, only patients with favorable performance status are eligible to receive these regimens.

The sponsor therefore considered a new concept of sequential GABRINOX treatment combining GEMBRAX followed by FOLFIRINOX, which should make it possible, by reducing toxicities, to increase the response rate and at the same time progression-free survival and median survival.

The sponsor performed a phase 1/2 study evaluating this GABRINOX protocol with the main objective of determining the maximum tolerated dose and increasing the response rate. Phase 2 is encouraging with a disease control rate and an objective response rate of 84.2% and 64.9% respectively, progression-free survival at 10.5 months and overall survival at 15.1 months as well as a more favorable safety profile compared to non-sequential treatments (less neutropenia 34.5%, febrile neutropenia 3.5% and neurotoxicity 5.2%).

These encouraging results led the investigator to propose a phase 2 study comparing the standard first-line treatment regimen FOLFIRINOX with the sequential regimen GABRINOX with the main objective of comparing efficacy in terms of objective response rate.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 75 on the date the consent is signed.
2. Histologically or cytologically proven metastatic pancreatic adenocarcinoma. The definitive diagnosis of pancreatic adenocarcinoma metastases will be made by integrating the histopathological data in the context of the radiological data.
3. One or more metastatic lesion (s) measurable (Recist 1.1) by Thoraco-Abdomino-Pelvic scanner (or hepatic MRI and Thoraco-Abdomino-Pelvic scanner not injected, if the patient is allergic to the product of contrast).
4. Previous treatment (including radiochemotherapy) for the non-metastatic disease authorized if a delay ≥ 6 months between the last treatment and the recurrence is respected.
5. WHO performance status ≤ 1
6. Uracilemia <16 ng / ml
7. Acceptable hematological assessment at inclusion (obtained within 14 days before the start of treatment) defined by: • Neutrophils ≥ 2 × 109 / L; • Platelets ≥ 100,000 / mm3 (100 × 109 / L); • Hemoglobin ≥ 9 g / dl.
8. Acceptable renal and hepatic function at inclusion (obtained within 14 days before the start of treatment) defined by: • AST and ALT ≤ 2.5 x upper limit of the norm (ULN), unless liver metastases are present in this case AST and ALT ≤ 5 × ULN is allowed; • Total bilirubin ≤ 1.5 x ULN; • Serum creatinine within the norm limits or calculated clearance ≥ 50ml / min for patients with a serum creatinine value above or below the norm values (clearance calculated by the CKD-EPI formula).
9. Calcemia AND magnesemia AND kalaemia ≥ LLN and ≤ 1.2 x ULN
10. If the patient is sexually active, he must agree to use contraception deemed adequate and appropriate by the investigator throughout the period of administration of the study drug and up to 6 months after discontinuation of treatment for women and for men.
11. Signature of consent before any procedure specific to the study.
12. Affiliated with the French national social security.

Exclusion Criteria:

1. Known brain metastasis.
2. Previous treatment with radiotherapy, surgery, chemotherapy or experimental therapy for the treatment of metastatic disease.
3. Major surgery, other than diagnostic surgery (that is, surgery done to obtain a diagnostic biopsy without organ harvesting), within 4 weeks of day 1 of study treatment.
4. Known Gilbert's syndrome or homozygous for know UGT1A1 * 28
5. Other concomitant cancer or history of cancer, except cervical cancer in situ treated, skin basal or squamous cell carcinoma, superficial bladder tumor (Ta, Tis, and T1) or a tumor with a good prognosis treated curatively without chemotherapy and without any sign of disease in the 3 years preceding inclusion.
6. Patients with high cardiovascular risk, including, but not limited to, coronary stent or myocardial infarction within the past 6 months.
7. Peripheral sensory neuropathy ≥ grade 2 at the time of inclusion.
8. ECG with a QTc interval greater than 450 ms for men and greater than 470 ms for women
9. Any other concomitant and unbalanced disease or serious disturbance that may interfere with the patient's participation in the study and his safety during the study (eg severe hepatic, renal, pulmonary, metabolic, or psychiatric disorders)
10. Allergy or intolerance to any study drug (gemcitabine, nab-paclitaxel, oxaliplatin, irinotecan, 5-FU) or any excipient (e.g., fructose) as described in the sections " contraindication or special warnings and precautions" or "prescribing information" of the summary of product characteristics indications.
11. Pregnant or breastfeeding women. Women of childbearing potential must have a negative pregnancy test (serum β-hCG) within 72 hours prior to inclusion.
12. Patients on vitamin K antagonists (e.g., Coumadin) (modifications to treatment may be required prior to inclusion).
13. Treatment with brivudine within 4 weeks before or after treatment with 5-fluorouracil (due to a potentially fatal interaction).
14. Active and uncontrolled bacterial, viral, or fungal infections requiring systemic treatment.
15. Active HIV infection, known hepatitis B or C infection.
16. History of peripheral arterial disease (e.g., claudication, Buerger's disease), chronic inflammatory bowel disease or rectal disease, pulmonary fibrosis or interstitial pneumonia.
17. Administration of a live attenuated vaccine within 10 days before inclusion and up to 6 months post-treatment.
18. Patient refusal or inability to comply with study procedures.
19. Inability to undergo follow-up for geographical, social, or psychological reasons.
20. Participation in another clinical trial involving an investigational product within the 30 days prior to inclusion.
21. Legal incapacity (patient under guardianship or guardianship).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From randomization to disease progression or death, up to 6 month
  To compare progression-free survival between the investigational treatment (Arm A) and the standard treatment (Arm B) in patients with metastatic 1st line pancreatic adenocarcinoma.
  Progression-free survival defined as the time between randomization and the onset of the 1st documented progression or death from any cause.
  Tumor progression is assessed according to the RECIST 1.1 criteria and by the centralized review.

SECONDARY OUTCOMES:
Tolerability of treatments | From randomization to 30 days after end of treatment, up to 13 month for Arm A and 7 month for Arm B
  Adverse events rate assessed according to the NCI-CTC AE V5.0 classification in application
Objective response rate | From randomization to the best response (complete or partial response) during treatment, up to 6 month
  Objective response rate (best response during treatment) defined as the percentage of complete or partial response. The tumor response is evaluated according to the RECIST 1.1 criteria.
Disease control rate | From randomization to the complete or partial response or stability, up to 6 month
  Disease control rate defined as the percentage of complete or partial response or stability.
  The tumor response is evaluated according to the RECIST 1.1 criteria.
Overall survival | From randomization to death, up to 2 years
  Overall survival defined as the time between randomization and the onset of death regardless of the cause.
Quality of life questionnaire -Core 30 (QLQ-C30) | At inclusion, then every 2 months up to 12 months then at 16 months, 20 months and 24 months (2 years)
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials. The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life questionnaire -PAN 26 | At inclusion, then every 2 months up to 12 months then at 16 months, 20 months and 24 months (2 years)
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life in patients with pancreatic cancer in clinical trials.
  The module comprises 26 questions assessing pain, dietary changes, jaundice, altered bowel habit, emotional problems related to pancreatic cancer, and other symptoms (cachexia, indigestion, flatulence, dry mouth, taste changes). The QLQ-PAN26 uses for the question 31 to 56 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much").
Collection of circulating tumor DNA (ctDNA) | At inclusion and when treatment is stopped (approximately 6 month)
  Establish a biological database for the analysis of biological predictive factors

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne PORTALES, MD, Study Chair — Institut de Cancérologie de Montpellier (ICM)
Locations (8):
- France (8):
  - CHU Grenoble, Grenoble, Auvergne-Rhône-Alpes
  - CHU St Etienne, Saint-Etienne, Auvergne-Rhône-Alpes
  - Institut GODINOT, Reims, Grand Est
  - CHU St Eloi, Montpellier, Herault
  - Institut régional du Cancer de Montpellier, Montpellier, Hérault
  - Centre Catalan d'Oncologie, Perpignan, Pyrénées-Orientales
  - CH de Perpignan, Perpignan, Pyrénées-Orientales
  - Centre Georges-François Leclerc, Dijon

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication and all sutdy documents can be share.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 years
Access Criteria: The data of the participants will be available on request and with a contract between the promoter and the applicant.
  The study protocol, the statistical analysis plan and the analytical code may also be the subject of data sharing under a transfer contract (GDPR-EU).

REFERENCES:
- [Background] Ferlay J, Partensky C, Bray F. More deaths from pancreatic cancer than breast cancer in the EU by 2017. Acta Oncol. 2016 Sep-Oct;55(9-10):1158-1160. doi: 10.1080/0284186X.2016.1197419. Epub 2016 Aug 23. PMID 27551890
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Sultana A, Smith CT, Cunningham D, Starling N, Neoptolemos JP, Ghaneh P. Meta-analyses of chemotherapy for locally advanced and metastatic pancreatic cancer. J Clin Oncol. 2007 Jun 20;25(18):2607-15. doi: 10.1200/JCO.2006.09.2551. PMID 17577041
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Derived] Portales F, Gourgou S, Fiess C, Salasc F, Assenat E, Ychou M. GABRINOX-2 protocol: a French, prospective, multicentre, randomised phase II trial evaluating gemcitabine/nab-paclitaxel followed by FOLFIRINOX versus FOLFIRINOX alone as first-line treatment for metastatic pancreatic cancer. BMJ Open. 2025 Aug 16;15(8):e104228. doi: 10.1136/bmjopen-2025-104228. PMID 40819868
- See also: Descriptive epidemiology of cancers in metropolitan France: incidence, survival and prevalence. Cowppli-Bony A, Colonna M, Ligier K, Jooste V, Defossez G, Monnereau A, et al. — https://linkinghub.elsevier.com/retrieve/pii/S0007455119300670